CLINICAL TRIAL: NCT00562471
Title: A Controlled Randomized Multicenter Study to Assess the Safety and Performance of Adhibit™ Adhesion Prevention Gel in Myomectomy Surgery
Brief Title: Safety and Efficacy Study of a Hydrogel, Applied Following Removal of Myomas During Gynecologic Surgery, Administered for the Prevention/Reduction of Postoperative Adhesion Formation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Angiotech Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADH-02-1; ADH-02-1.1; ADH-02-1.2; ADH-02-1.3
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Myoma
Keywords: adhesions; gynecologic surgery; laparoscopy; laparotomy; polyethylene glycol; hydrogel; Adhesions following gynecologic surgery to remove myomas
MeSH Terms: conditions — Myoma; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Adhesion Prevention Gel Arm
  Interventions: Other: Adhibit Adhesion Prevention Gel
- 2 (Other): Standard of Care Comparator Arm (standard of care for post-operative adhesion prevention included irrigation of tissues and lavage of all fluids with Ringers Lactate solution following surgery and 300 to 500mL of solultion left in the pelvic cavity immediately prior to wound closure)
  Interventions: Other: Standard of Care Comparator

INTERVENTIONS:
Other: Adhibit Adhesion Prevention Gel — A resorbable hydrogel, which adheres to itself and the tissues it contacts, is approved for use in sealing vascular reconstructions. The hydrogel is formed when two synthetic derivatized polyethylene glycol (PEG) polymers are mixed together and applied to tissue. Using a gas-assisted delivery device, the hydrogel is sprayed over all myomectomy suture lines and all surgically treated areas during the myomectomy surgery. The hydrogel is totally resorbed within 30 days post-application.
  Other Names: CoSeal Surgical Sealant; CoSeal Adhesion Prevention Gel
  Arms: 1
Other: Standard of Care Comparator — standard of care for post-operative adhesion prevention included irrigation of tissues and lavage of all fluids with Ringers Lactate solution following surgery and 300 to 500mL of solultion left in the pelvic cavity immediately prior to wound closure
  Arms: 2

SUMMARY:
The purpose of this study was to determine whether the adhesion prevention gel was safe to use, and was effective for the prevention/reduction of adhesion formation that typically occurs following gynecological surgery to remove myomas

DETAILED DESCRIPTION:
Postoperative adhesions are a common medical complication of gynecologic and pelvic surgeries, and are frequently associated with chronic or recurrent pelvic pain, intestinal obstruction and infertility. This randomized, controlled, multicenter, clinical study was designed to evaluate the safety and performance of Adhibit™ Adhesion Prevention Gel versus the standard of care for the reduction of postoperative adhesions in subjects undergoing myomectomy via laparotomy or laparoscopy. Subjects were scheduled to return within 6-8 weeks after the initial surgical procedure. At that time, a second-look laparoscopy was performed for postoperative adhesion assessment. Adhesions were graded using a modified American Fertility Society (mAFS) scoring method.

ELIGIBILITY:
Inclusion Criteria:

Preoperatively, subjects must have had:

* Been scheduled for myomectomy via laparotomy or laparoscopy.
* Agreed to a second-look laparoscopic procedure to assess and lyse any adhesions formed at 6 to 8 weeks following myomectomy.
* Been >=18 years of age.
* Provided voluntary written informed consent.
* Been willing to comply with all aspects of the treatment and evaluation schedule.

Intra-operatively, subjects must have had:

* Had at least one 2 cm incision length on posterior uterine surface, which may include the fundal surface.

Exclusion Criteria:

Preoperatively, subjects must not have had:

* Been pregnant.
* Had a pelvic malignancy.
* Had acute pelvic inflammatory disease.
* Had an immune compromised condition.
* Been a participant in another clinical research study which the investigator believed could interfere with the purpose of this study.
* Been given corticosteroids intra-operatively or during the course of the postoperative study follow up.

Intra-operatively, subjects must not have had:

* Had a pelvic malignancy.
* Had a pelvic or abdominal infection.
* Had acute pelvic inflammatory disease.
* Received any adhesion prevention adjuvants or barriers, or peritoneal instillates containing corticosteroids, NSAIDs, or Dextran.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-07; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
modified American Fertility Society (mAFS) score at the posterior uterus | 6-8 weeks following primary myomectomy surgery

SECONDARY OUTCOMES:
adhesion extent and tenacity scores at the posterior uterus | 6-8 weeks following primary myomectomy surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte METTLE, MD, PhD, Principal Investigator — Univ. Clinics of Schleswig-Holstein
Locations (6):
- St. Joseph's Health Centre, Toronto, Ontario, Canada
- Germany (4):
  - Klinik für Minimal Invasive Chirurgie, Berlin
  - Universitätsklinikum Giessen, Giessen
  - Univ. Clinics of Schleswig-Holstein, Kiel
  - Bethesda Krankenhaus Wupperta, Wuppertal
- St. Elizabeth Hospital, Curaçao, Netherlands Antilles

REFERENCES:
- [Derived] Mettler L, Hucke J, Bojahr B, Tinneberg HR, Leyland N, Avelar R. A safety and efficacy study of a resorbable hydrogel for reduction of post-operative adhesions following myomectomy. Hum Reprod. 2008 May;23(5):1093-100. doi: 10.1093/humrep/den080. Epub 2008 Mar 17. PMID 18346996